CLINICAL TRIAL: NCT06572566
Title: Study on the Mechanism of Action of Chemical Category 1 Innovative Drug GMDTC on Neuropsychiatric Behavior in Cadmium-exposed People
Brief Title: Study on Neuropsychiatric Behavior in Cadmium-exposed People
Status: Recruiting | Type: Observational
Sponsor: Jianersheng (Zhuhai) Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JianerShengPharmaNI
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cadmium Exceeds the Standard
Keywords: cadmium; Cadmium exceeds the standard; neuropsychiatric behavior; neuroimaging; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cadmium exceeding standard group: The urine cadmium level exceeding 5 μg/g creatinine for two consecutive times.
  Interventions: Other: Non-invasive examination and assessment.
- healthy control group: Urine cadmium ≤ 5 μg/g creatinine.
  Interventions: Other: Non-invasive examination and assessment.

INTERVENTIONS:
Other: Non-invasive examination and assessment. — 1) Test the blood and urine components of all subjects to evaluate the damage to kidney function caused by excessive cadmium. 2) Conduct MRI examinations on all subjects to evaluate changes in brain functional connectivity, metabolism, and structure after excessive cadmium exposure. 3) Conduct bone density examinations on all subjects to evaluate changes in bone density after excessive cadmium exposure. (3) Clinical psychiatric assessment: All subjects will be assessed on their mental and psychological conditions such as pain, cognitive function, depression, anxiety, mania, sleep quality, and suicide risk.

SUMMARY:
This study hypothesized that excessive cadmium is related to clinical pain, depression, and cognitive impairment, and that related indicators will improve after cadmium is eliminated.

DETAILED DESCRIPTION:
This study will combine the research progress of the innovative drug GMDTC, the mechanism of nerve damage caused by Cd2+ disrupting Ca2+ homeostasis, imaging technology and analysis methods, and the basis of our previous research work to explore the effect of the chemical Class 1 innovative drug GMDTC on the neuropsychiatric behavior of people with excessive cadmium. mechanism of action. This study is not limited to the study of the mechanism of neurotoxicity after Cd2+ deposition. It will also clarify the clinical efficacy of the innovative drug GMDTC in removing Cd2+ deposition in the brain and reducing damage, which is expected to open up new avenues for the treatment of cadmium neurotoxicity. This study hypothesized that excessive cadmium is related to clinical pain, depression, and cognitive impairment, and that related indicators will improve after cadmium is eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, both men and women are welcome
* The weight of male subjects is ≥50.0 kg, the weight of female subjects is ≥45.0 kg, and the body mass index (BMI) is between 19 ~ 26 kg/m2, including the critical value
* Urinary cadmium >5 μmol/mol creatinine for 2 consecutive days (creatinine content is ≥0.3 μg/L and ≤3 μg/L)
* Right-handed
* Voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

* Combined with other neurodevelopmental problems (such as autism), organic brain mental disorders (such as Alzheimer's disease, Parkinson's disease, etc.) and organic brain diseases (such as cerebral hemorrhage, infarction, etc.) that meet the DSM-5 diagnostic criteria )
* Those who have suffered from or are currently suffering from any serious clinical diseases that pose safety risks such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities
* Continuous use of high-dose neuroleptics in the past 3 months (high-dose: daily dosage of benzodiazepines ≥ 4 mg lorazepam equivalent; long-term: the total duration of use is at least 60 days)
* Have contraindications for MRI or bone density examination (pacemaker or defibrillator, artificial heart valve, clothing containing fluorescein, iron, etc.)
* Pregnant and lactating women
* Those who cannot tolerate venipuncture and/or have a history of fainting from blood or needles
* Those with eGFR <30 mL/min/1.73 m2 during screening (eGFR is calculated using the Cockcroft-Gault formula: eGFR(mL/min/1.73m2) = (140-age)*weight (kg)/[0.818*Cr(μmol/L )]*0.85(female))

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were recruited from the cadmium-excessive group at the Hunan Provincial Occupational Disease Prevention and Control Hospital from January 2024 to June 2024, and healthy volunteers were recruited from the outpatient clinic. It is planned to include 42 cases of people with excessive cadmium and 42 cases of healthy people.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cadmium load | Baseline, after 2 weeks, after 6 weeks
  To comprehensively assess the urinary cadmium levels in volunteers, blood cadmium and urinary cadmium levels were measured at different time points.
McGill Pain Questionnaire Short Form (MPQ) | Baseline, after 2 weeks, after 6 weeks
  Pain was measured through the McGill Pain Questionnaire Short Form (MPQ)，The scale will include the unabbreviated scale title, the minimum and maximum values, and higher scores mean a worse outcome.
MATRICS Consensus Cognitive Battery (MCCB) | Baseline, after 2 weeks, after 6 weeks
  The internationally recognized MATRICS Consensus Cognitive Battery (MCCB) for objective assessment of cognitive function.Cognitive scores for all individuals will be calculated using the MCCB software, yielding corrected scores for each test as well as an overall cognitive score.
The Hamilton Depression Rating Scale (HAMD) | Baseline, after 2 weeks, after 6 weeks
  mental and psychological status was assessed with the Hamilton Depression Rating Scale (HAMD).The scale will include the unabbreviated scale title, the minimum and maximum values, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
One of the early indicators of kidney injury--β2-MG | Baseline, after 2 weeks, after 6 weeks
  β2-microglobulin(β2-MG).Clinically, the measurement of β2-MG concentration in urine provides an early, reliable, and sensitive indicator for assessing renal function and diagnosing cadmium toxicity.
Hamilton Anxiety Scale（HAMA） | Baseline, after 2 weeks, after 6 weeks
  The HAMA scale will be used to assess the anxiety levels of volunteers, with higher scores indicating more severe anxiety.
One of the early indicators of kidney injury--NAG | Baseline, after 2 weeks, after 6 weeks
  N-acetyl-β-D-glucosaminidase,NAG. Urinary N-acetyl-beta-D-glucosaminidase (NAG) activity is one of the sensitive and specific indicators for renal tubular lesions and can serve as an early diagnostic marker for tubular damage, even providing earlier predictive value than urinary albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Pei, Principal Investigator — Hunan Occupational Disease Prevention and Control Institute
Locations (1):
- Hunan Occupational Disease Prevention and Control Institute, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemens S, Aarts MG, Thomine S, Verbruggen N. Plant science: the key to preventing slow cadmium poisoning. Trends Plant Sci. 2013 Feb;18(2):92-9. doi: 10.1016/j.tplants.2012.08.003. Epub 2012 Sep 12. PMID 22981394
- [Background] Deng D, Xu C, Sun P, Wu J, Yan C, Hu M, Yan N. Crystal structure of the human glucose transporter GLUT1. Nature. 2014 Jun 5;510(7503):121-5. doi: 10.1038/nature13306. Epub 2014 May 18. PMID 24847886
- [Background] Mergenthaler P, Lindauer U, Dienel GA, Meisel A. Sugar for the brain: the role of glucose in physiological and pathological brain function. Trends Neurosci. 2013 Oct;36(10):587-97. doi: 10.1016/j.tins.2013.07.001. Epub 2013 Aug 20. PMID 23968694